CLINICAL TRIAL: NCT00608127
Title: A Single - Arm Open - Label Study to Evaluate the Safety, Tolerability and Short Term Efficacy of Extracorporeal Specific Immunoadsorption LupusorbTM Columns for the Treatment of Systemic Lupus Erythematosus (SLE) Patients
Brief Title: Study to Evaluate the Safety, Tolerability and Short Term Efficacy of Extracorporeal Specific Immunoadsorption LupusorbTM Columns for the Treatment of Systemic Lupus Erythematosus (SLE) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Verto LTD (Industry)
Responsible Party: Dr. Anat Scheiman, Hadassah Medical Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUP-001-ISR
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single arm open label
  Interventions: Device: LupusorbTM

INTERVENTIONS:
Device: LupusorbTM — Single treatment

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a chronic, autoimmune, inflammatory disease primarily affecting women of childbearing age, and associated with severe morbidity and mortality of its victims. The existing therapy, however, is not specific and its inevitable side effects may themselves be fatal. Therefore, it is a widely recognized need for, and it would be highly advantageous to have a safe, specific rapidly effective and well-defined treatment of SLE, devoid of the disadvantages.

We have shown that VRT101 a peptide present in the extracellular laminin is a target for pathogenic lupus autoantibodies. Using this peptide we have developed the LupusorbTM - an immune-adsorption column which specifically binds pathogenic antibodies from monoclonal cultures as well as from patients' plasma. The investigational product named LupusorbTM Column is a sterile medical device for single use and can be classified into category IIb (synthetic ligands, peptides) according to Annex IX of the European Medical Device Directive 42/93/EEC.

The proposed study, a pilot non-randomized open label study, will test the safety, Tolerability and short term efficacy of a single immunoadsorption procedure in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants, either male or female are at least 18 years of age at entry.
2. Have diagnosed documented SLE, determined at least by 4 criteria as defined by the American Rheumatism Association ARA
3. Active SLE disease with a SLEDAI score greater than 3
4. Serum anti-VRT101 at least 0.4 O.D.
5. Be willing and able to comply with the protocol for the duration of the study.
6. Participant understands the nature of the procedure and provides written informed consent prior to any study procedure.
7. If female, must be neither pregnant nor breast-feeding and must lack childbearing potential for the duration of the study.

Exclusion Criteria:

Subjects will be excluded from the study if ANY of the following conditions are present:

1. Patient has Severe proliferative lupus nephritis:

   1. Rapidly progressive glomerulonephritis (doubling of serum creatinine during last 3 months); or
   2. Severe impairment of renal function Cr more than 2.5 mg/dL
2. Patient Begin immunosuppressive therapy recently:

   1. Beginning treatment with azathioprine, mycophenolic acid, cyclosporine or methotrexate within 4 weeks.
   2. Cyclophosphamide-an IV pulse within the last 3 months
   3. Pulse therapy with glucocorticoids during the 4 weeks before study entry.
   4. Patient is in on another experimental therapy.
3. Patient suffers an active or chronic infection.
4. If female, reports pregnancy, breast-feeding (or inadequate birth control)
5. Confounding medical illness that in the judgment of investigators would pose.

   Added risk for study participants such as:
   1. Unstable coronary artery disease, cardiomyopathy or dysrhythmia requiring therapy
   2. Hematologic disease (Hb < 7 G/dL, platelets < 50,000/dL or WBC < 2,000/dL).
   3. Bleeding tendency
   4. Hypogammaglobulinemia (Serum IgG< 500mg/dL)
6. Participation in another clinical trial within 2 months prior to start of this study.
7. Subject unwilling or unable to comply with the requirements of the protocol.
8. Any condition that the investigator feels would interfere with trial participation and evaluation of the results.
9. Subject unwilling and unable to provide inform consent.
10. Subjects receiving ACE inhibitors treatment 7 days prior to plasmapheresis procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-05 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Safety assessment- Patient's physical examination, vital signs (HR, BP, RR, Rhythm status), lab tests- hematology, CBC & blood biochemistry, Serology panel, anti VRT101 levels, liver and kidney function, urinalysis and SLE serological markers. | Within 2 months

SECONDARY OUTCOMES:
Efficacy assessment- SLE severity, CBC with differential, ESR, CRP, Blood biochemistry: Serum albumin, Serum Igs, Serology panel: ANA, direct Coomb's; C3, C4, anti-DNA and Serum anti-VRT 101 level and SF 36 Health questionnaire. | within 2 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Ein- Kerem, Jerusalem, Israel